CLINICAL TRIAL: NCT01640093
Title: A Single-Dose, Open-Label, Randomized, 4-Way Crossover Study to Assess the Relative Bioavailability of 3 New Abiraterone Acetate Tablet Formulations With Respect to the Current Commercial Abiraterone Acetate Tablet Under Fasted Conditions in Healthy Male Subjects
Brief Title: A Comparative Study of Bioavailability of 3 New Abiraterone Acetate Tablets With Current Commercial Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100859; 212082PCR1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Bioavailability; Pharmacokinetics; Abiraterone acetate; Abiraterone
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment B (Experimental): Abiraterone acetate (500 mg), 2 coated, reformulated tablets.
  Interventions: Drug: Abiraterone acetate, 500 mg (coated, reformulated tablet)
- Treatment C (Experimental): Abiraterone acetate (250 mg), 4 coated, reformulated tablets.
  Interventions: Drug: Abiraterone acetate, 250 mg (coated, reformulated tablet)
- Treatment D (Experimental): Abiraterone acetate (500 mg), 2 coated, reformulated tablets, showing slower in vitro dissolution.
  Interventions: Drug: Abiraterone acetate, 500 mg (coated tablet, slower in vitro dissolution)
- Treatment A (Active Comparator): Abiraterone acetate (250 mg), 4 uncoated, current commercial tablets.
  Interventions: Drug: Abiraterone acetate, 250 mg (uncoated, current commercial tablet)

INTERVENTIONS:
Drug: Abiraterone acetate, 250 mg (uncoated, current commercial tablet) — Type=exact number, unit=mg, number=250, form=tablet, route=oral. Administered once under fasted conditions.
  Other Names: ZYTIGA
  Arms: Treatment A
Drug: Abiraterone acetate, 500 mg (coated, reformulated tablet) — Type=exact number, unit=mg, number=500, form=tablet, route=oral. Administered once under fasted conditions.
  Other Names: ZYTIGA
  Arms: Treatment B
Drug: Abiraterone acetate, 250 mg (coated, reformulated tablet) — Type=exact number, unit=mg, number=250, form=tablet, route=oral. Administered once under fasted conditions.
  Other Names: ZYTIGA
  Arms: Treatment C
Drug: Abiraterone acetate, 500 mg (coated tablet, slower in vitro dissolution) — Type=exact number, unit=mg, number=500, form=tablet, route=oral. Administered once under fasted conditions.
  Other Names: ZYTIGA
  Arms: Treatment D

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (what the body does to the medication) and relative bioavailability of 3 newly developed abiraterone acetate tablet formulations compared with the current commercial abiraterone acetate tablet formulation in healthy male participants, under fasted conditions, at a single dose of 1000 mg.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), single-center, 4-way crossover study (method used to switch participants from one treatment arm to another in a clinical trial) of a single dose of abiraterone acetate (1000 mg). The study will consist of 3 phases including screening phase (of 21 days), an open-label treatment phase consisting of 4 single-dose treatment periods, and follow-up phase. All participants will be randomly assigned to 1 of 4 possible treatment sequences to ensure that they receive all of the following treatments, one in each period. The 4 sequences are as follows: Sequence 1: Treatment A, D, B, and C; Sequence 2: Treatment B, A, C, and D; Sequence 3: Treatment C, B, D, and A; and Sequence 4: Treatment D, C, A, and B. After a washout period of 7 days, follow-up phase will occur between 5 to 7 days after the last study procedure. The duration of participation in the study for each participant is from 47 days to a maximum of 68 days (including screening). Pharmacokinetics will be measured by collection of blood samples. Participants will be confined to the study center until completion of the 96 hour pharmacokinetic assessments on Day 5 of each treatment period. Safety evaluations for adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examinations will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have body weight not less than 50 kg
* Must be a non-smoker, and has no history of smoking or use of nicotine-containing substances within the previous 2 months
* Must have blood pressure between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* Must have a 12-lead electrocardiogram consistent with normal cardiac conduction and function
* Must agree to use an adequate contraception method as deemed appropriate by the investigator and to not donate sperm during the study for 3 months after receiving the last dose of study medication

Exclusion Criteria:

* History of or current clinically significant medical illness including cardiac arrhythmias or other cardiac disease that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology or urinalysis (at screening)
* Clinically significant abnormal physical examination vital signs or 12-lead electrocardiogram (at screening)
* Usage of any prescription or nonprescription medication, except for acetaminophen, and oral contraceptives and hormonal replacement therapy within 14 days before the first dose of the study medication is scheduled
* Unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study medication)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of abiraterone in coated, reformulated tablet compared to abiraterone in uncoated, current commercial tablet | For each period: Predose, 15 min, 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours, and at 96 hours
  Pharmacokinetic parameter Cmax of abiraterone (coated, reformulated tablet and uncoated, current commercial tablet) will be measured when abiraterone acetate is administered as a single oral 1000-mg dose.
Area under the plasma concentration versus time curve (AUC) of abiraterone in coated, reformulated tablet compared to abiraterone in uncoated, current commercial tablet | For each period: Predose, 15 min, 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours, and at 96 hours
  Pharmacokinetic parameter AUC of abiraterone (coated, reformulated tablet and uncoated, current commercial tablet) will be measured when abiraterone acetate is administered as a single oral 1000-mg dose.

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 68 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States